CLINICAL TRIAL: NCT02453321
Title: A Comparison Between Continuous Selective Femoral Blocks and Continuous Adductor Canal Blocks at Mid-Thigh in Total Knee Arthroplasty: What is the Best Method to Optimize Functional Achievement and Analgesia in Early Rehabilitation?
Brief Title: Continuous Adductor Canal Blocks Vs. Low Dose Femoral Nerve Blocks For Early Rehabilitation After Total Knee Arthroplasty
Acronym: FemVsACB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kevin King, DO (Other)
Responsible Party: Sponsor-Investigator, Kevin King, DO, Clinical Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO13110481
Record Dates: First submitted 2015-04-24; First posted 2015-05-25 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Pain, Postoperative; Total Knee Arthroplasty (TKA)
Keywords: Continuous Femoral Nerve Block; Continuous Adductor Canal Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Nerve Block; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cont. Femoral Block - Low Dose Group (Active Comparator): Arm is named by the intervention the group receives. Continuous Femoral Block - Low Dose. The Block/catheter is placed about 5cm below groin at ultrasonographic apex of femoral triangle. Rate of 2ml/hr of bupivacaine 0.0625% until morning of POD#2.
  Interventions: Procedure: Continuous Femoral Nerve Block; Procedure: Continuous Sciatic Nerve Block; Drug: Bupivacaine
- Cont. Femoral Block - Higher Dose (Experimental): Place the CPNB in same manner as low-dose group, but rate will be 4ml/hr. Hypothesis is that this group may experience better pain control, but likely will have more dense motor blockade of thigh and less participation in physical therapy
  Interventions: Procedure: Continuous Femoral Nerve Block; Procedure: Continuous Sciatic Nerve Block; Drug: Bupivacaine
- Continuous Adductor Canal (Experimental): Placed at mid-thigh in proximal adductor canal near femoral artery with a bupivacaine infusion rate of 4ml/hr. Hypothesis is that this group may experience less motor blockade of thigh but may have more pain than the femoral nerve groups.
  Interventions: Procedure: Nerve Block, Continuous Adductor Canal; Procedure: Continuous Sciatic Nerve Block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Continuous Femoral Nerve Block — A 27g plastic catheter placed below the inguinal crease to perform a conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Other Names: Continuous Nerve Block, Femoral; Continuous Peripheral Nerve Block
  Arms: Cont. Femoral Block - Higher Dose; Cont. Femoral Block - Low Dose Group
Procedure: Nerve Block, Continuous Adductor Canal — A 27g plastic catheter placed on the anterior medial thigh midway between the groin and knee to provide a local anesthetic conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Other Names: Continuous Nerve Block, Adductor Canal; Continuous Peripheral Nerve Block, Adductor Canal
  Arms: Continuous Adductor Canal
Procedure: Continuous Sciatic Nerve Block — A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Other Names: Nerve Block, Sciatic Continuous
Drug: Bupivacaine — The concentration of the continuous infusion of bupivacaine though the peripheral nerve catheters will be 0.0625% for the femoral and adductor canal blocks and the concentration for the sciatic continuous catheter will be 0.03%.

SUMMARY:
Recently, several articles have suggested or reported that Adductor Canal Blocks (ACBs) offer adequate or equal analgesia and may promote better performance in early rehabilitation following Total Knee Arthroplasty (TKA) when compared to the more commonly used Femoral Nerve Block (FNB). A common feature of these studies has been the use of moderate to high concentration local anesthetics (e.g. 0.2% or 0.5% Ropivacaine respectively) which when injected by a large motor nerve will inevitably cause weakness. However, the practice at our institution has long been a continuous femoral nerve block (CFNB) with a lower concentration local anesthetic (0.0625% Bupivacaine). Over the past several years the investigators have performed several thousand CFNBs using this technique which has offered the advantage of minimal motor weakness and adequate analgesia.

The primary goal of this study is to determine if our established practice of using a low concentration continuous FNB inserted about 5cm caudal to the groin crease (the apex of the femoral triangle) using a low infusion rate of 2ml/hr is comparable to the emerging practice of inserting a Continuous Peripheral Nerve Block (CPNB) in the anatomic adductor canal (AC) - infusing at 4ml/hr. A secondary goal is to study the effect of cumulative volume of local anesthetic infused through a FNB when at a rate of 2ml/hr compared to a rate of 4ml/hr in the 48-hour postoperative period.

Definitions of the location of the adductor canal are debated heavily in literature, but they seem to agree that the middle 1/3 of the thigh contains the proximal AC while the distal 1/3 of the thigh contains the adductor hiatus - the terminal end of the AC. Our study will require placement of the continuous ACB no more distal than 20cm cephalad to the superior pole of the patella due to placement prior to surgery and the need to keep the dressing out of the operative field. The CACB catheter will also not be placed any more proximal than 20cm distal to the ASIS. In addition to other exclusion criteria, these measurements will create an exclusion for patients with an iliac-to-patella distance less than 40cm. Iliac to Patella distance (IPD) will be measured at the pre-operative interview on the day of surgery with a measuring tape. External palpable landmarks of the Anterior superior iliac spine and the superior pole of the patella will be used.

The primary outcome is based upon the ability to perform rehabilitation exercises postoperatively to the extent that criteria for discharge can be met. The primary outcome measured is the time at which a patient gains the ability to successfully perform a 75-feet unassisted walk. On the Day of Surgery (DOS), prior to any walking attempt, a secondary outcome measure will be to perform a 5-second sustained straight leg raise. Other secondary outcomes will be the number of days admitted prior to discharge, and average pain scores on DOS, Postoperative Day (POD) #1, and POD#2. The Day of discharge will also be used as a secondary outcome. Earlier discharge is becoming a goal of almost all healthcare systems to minimize costs.

DETAILED DESCRIPTION:
The three arms are as follows:

1. The control group; Continuous Femoral Nerve Block - Low Dose (CFNB-LD) will be patients randomized to our standard therapy comprised of a low dose/concentration Continuous Femoral Nerve Block inserted approximately 5cm distal to the groin crease with a rate of 2ml/hr.
2. Higher dose (HD) CFNB; - block placed in same location as CFNB-LD but with a higher dose rate of 4ml/hr. This higher rate could afford more pain control but may cause more quadriceps or hip flexor weakness.
3. Continuous Adductor Canal Block (CACB) group will have a catheter inserted 20-30cm proximal to the superior pole of the patella, and an infusion rate of 4ml/hr, but with similar dressing to make it appear like those in group 1 and 2.

Acute Pain/Regional anesthesiologists and fellows will be performing all research procedures in the same locations that the investigators routinely perform regional nerve blocks: our preoperative holding area adjacent to the operating room suites at University of Pittsburgh Medical Center (UPMC) - Passavant.

All three groups have a set rate that will not increase. There also will be no bolus orders given on the floors, however IV and PO medications will be available to decrease discomfort. These medications are ordered to be given upon request (PRN); upon patient request. Down-regulation of doses will also not be allowed as that would cause uncertainty as to which regimen may contribute most to postoperative weakness. The only adjustment allowed will be to turn off the nerve block infusion completely on POD #1 if a dense motor block of the quadriceps or iliopsoas (hip flexor) exists, as this condition does not facilitate participation in rehabilitation exercises. The frequency of early-removal of nerve block will be recorded for all three groups.

CFNB groups Continuous Femoral Nerve Block placement: The skin of the right or left groin will be sterilized and draped under sterile conditions, the femoral nerve will be identified using ultrasound just below the inguinal crease and the local anesthetic will be infiltrated subcutaneously. The needle is inserted at the lateral edge of the probe and directed toward the nerve using ultrasound assistance. When in proximity of the nerve, 15ml of 0.2% ropivacaine will be injected through the needle with repeat aspiration every 5 ml. The nerve block catheter will be placed 3-5 cm past the needle tip and secured with steri strips and bio-occlusive dressing.

CACB group Continuous Adductor Canal Block placement: The distance from the ASIS to the superior pole of the patella will be measured and the distance recorded. This Iliac-to-Patella distance (IPD) will be divided into proximal and distal halves, and the halfway point marked. The length of the IPD will need to be a minimum of 40cm for inclusion. The insertion site will need to be 20cm proximal to the superior pole of the patella and at least 20ml distal to the ASIS. The attending anesthesiologist / acute pain attending either perform or supervise regional anesthesia fellows to place the CACB no more proximal than the halfway mark of the IPD. For example, if a patient has an IPD of 50cm, the halfway mark will be at 25cm and this would be the site of insertion as it would be within the anatomic adductor canal and would be adequately removed from the surgical site. The skin of the right or left anterior-medial thigh will be sterilized and draped under sterile conditions. The sartorius muscle and femoral artery will be identified by an ultrasound at the marked IPD-halfway-mark. There, local anesthetic will be infiltrated subcutaneously. The needle is inserted in the direction of the hyperechoic nerve and the hypoechoic femoral artery using ultrasound assistance. When the needle tip is deep to the sartorius and in proximity of the artery, 15ml of 0.2% ropivacaine will be injected through the needle with repeat aspiration every 5 ml. The nerve catheter will be placed 3-5 cm past the needle tip and secured with steri-strips and bio-occlusive dressing. The CACB rate will be 4ml/hr of bupivacaine 0.0625%.

By design, Observers should only be aware of a singular kind of patient; those with CPNBs.

The dressing of the cACB will be very similar to the CFNB and the standard yellow connector piece will be secured to the skin with bio-occlusive covering, and the location will be at level of the anterior superior iliac spine (ASIS). This standardized dressing will serve to aid in blinding the observers as to which kind of continuous block the patient received. Labeling of the catheter and dressing will not differ. The nerve block billing record will contain the information on the particular approach used.

Sciatic nerve block placement: the corresponding right or left gluteal area will be sterilized and draped under sterile conditions, the sciatic nerve will be identified by an ultrasound in the lower gluteal region where a local anesthetic will be infiltrated subcutaneously. A trans-gluteal approach will be used to inject normal saline through the needle to assist catheter placement; the catheter will be introduced for 3-5 cm past the needle tip and secured with steri strips and tegaderm. No local anesthetic will be administered until the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent to regional anesthesia and having primary total knee arthroplasty/replacement

Exclusion Criteria:

* Body-Mass Index >40
* Iliac to Patella Distance (IPD) <40cm
* Pre-existing quadriceps weakness of involved surgical side Chronic opioid use (if using opioids within 4 weeks of surgery: excluded)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waters Jonathan, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center - Passavant Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting for Total Knee Arthroplasty (TKA) at University of Pittsburgh Medical Center (UPMC) - Passavant Hospital were approached on the day of surgery, but some were called the day prior to surgery.
Pre-assignment Details: No patients were enrolled but excluded prior to assignment to a randomized group.
Groups:
- Cont. Femoral Block - Low Dose Group: Continuous Femoral Block - Low Dose Intervention Group. The Block/catheter is placed about 5cm below groin at ultrasonographic apex of femoral triangle. Rate of 2ml/hr of bupivacaine 0.0625% until morning of Postoperative Day (POD) #2.
  Continuous Femoral Nerve Block: A 27g plastic catheter placed below the inguinal crease to perform a conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupi
- Cont. Femoral Block - Higher Dose: Place the Continuous Peripheral Nerve Block (CPNB) in same manner as low-dose group, with increased rate of 4ml/hr. Hypothesis is that this group may experience better pain control, but more motor blockade of thigh and less participation in physical therapy is likely.
  Continuous Femoral Nerve Block: A 27g plastic catheter placed below the inguinal crease to perform blockade of the sensory components of the femoral nerve to decrease pain in the knee after TKA.
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupivacaine tho
- Continuous Adductor Canal: Placed at mid-thigh in proximal adductor canal near femoral artery with a bupivacaine infusion rate of 4ml/hr. Hypothesis: This group may experience less motor blockade of thigh but may have more pain than the femoral nerve groups.
  Nerve Block, Continuous Adductor Canal: A 27g plastic catheter placed on the anterior medial thigh midway between the groin and knee to provide a local anesthetic conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: T
Period: Overall Study
Arm/Group | Cont. Femoral Block - Low Dose Group | Cont. Femoral Block - Higher Dose | Continuous Adductor Canal
Started | 20 | 21 | 21
Completed | 19 | 19 | 19
Not Completed | 1 | 2 | 2
Not completed — Weakness | 1 | 1 | 2
Not completed — Deep Venous Thrombosis | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cont. Femoral Block - Low Dose Group: Arm is named by the intervention received... Continuous Femoral Block - Low Dose. The Block/catheter is placed about 5cm below groin at ultrasonographic apex of femoral triangle. Rate of 2ml/hr of bupivacaine 0.0625% until morning of POD#2.
  Continuous Femoral Nerve Block: A 27g plastic catheter placed below the inguinal crease intended to block the sensory nerves to decrease pain in the knee after TKA.
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It is only dosed postoperatively after verifying sciatic nerve function is intact. The infusion is 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the infusions of bupivacaine in peripheral nerve catheters will be 0.0625% for the femoral and adductor canal, and
- Cont. Femoral Block - Higher Dose: Place the CPNB in same manner as low-dose group, but rate will be 4ml/hr. Hypothesis is that this group may experience better pain control, but likely will have more dense motor blockade of thigh and less participation in physical therapy
  Continuous Femoral Nerve Block: A 27g plastic catheter inserted below the inguinal crease to cause conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupivacaine tho
- Continuous Adductor Canal: Placed at mid-thigh in proximal adductor canal near femoral artery with a bupivacaine infusion rate of 4ml/hr. Hypothesis is that this group may experience less motor blockade of thigh but may have more pain than the femoral nerve groups.
  Nerve Block, Continuous Adductor Canal: A 27g plastic catheter placed on the antero-medial thigh midway between the groin and knee to provide a local anesthetic conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: T
- Total: Total of all reporting groups
Arm/Group | Cont. Femoral Block - Low Dose Group | Cont. Femoral Block - Higher Dose | Continuous Adductor Canal | Total
Number analyzed (Participants) | 20 | 21 | 21 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 12 | 13 | 13 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (5.5) | 67.0 (5.1) | 66.5 (6.8) | 66.2 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 8 | 33
  Male | 10 | 6 | 13 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 21 | 62

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Physical Therapy Discharge Criteria as Measured by 75-feet Walk Test. {Number of Hours After Conclusion of Surgery}
Description: Ability to walk 75 feet if performed on POD#2 is usually considered the main criterion for discharge at UPMC Passavant. The patient is accompanied/supervised by physical therapist using a walker but without active intervention by therapist, unless necessary. The earliest day on which the patient achieves the 75-feet unassisted walk will be recorded for comparison among the arms/groups.
Time Frame: Participants will be followed for the duration of hospital stay, an average of 4 days
Measure: Median (Inter-Quartile Range); unit: Hours
Groups:
- Cont. Femoral Block - Low Dose Group: Arm is named by the intervention received.. Continuous Femoral Block - Low Dose. The Block/catheter is placed about 5cm below groin at ultrasonographic apex of femoral triangle. Rate of 2ml/hr of bupivacaine 0.0625% until morning of POD#2.
  Continuous Femoral Nerve Block: A 27g plastic catheter placed below the inguinal crease to perform a conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupi
- Cont. Femoral Block - Higher Dose: Place the CPNB in same manner as low-dose group, but rate to be 4ml/hr. Hypothesis is that this group may experience better pain control, but likely will have more dense motor blockade of thigh and less participation in physical therapy
  Continuous Femoral Nerve Block: A 27g plastic catheter placed below the inguinal crease to perform a conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupivacaine tho
- Continuous Adductor Canal: Placed at mid-thigh in proximal adductor canal near femoral artery with a bupivacaine infusion rate of 4ml/hr. Hypothesis is that this group may experience less motor blockade of thigh but may have more pain than the femoral nerve groups.
  Nerve Block, Continuous Adductor Canal: A 27g plastic catheter placed on the antero- medial thigh midway between the groin and knee to provide a local anesthetic conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: T
Arm/Group | Cont. Femoral Block - Low Dose Group | Cont. Femoral Block - Higher Dose | Continuous Adductor Canal
Number analyzed (Participants) | 19 | 19 | 19
Hours | 67.3 [38.9 to 70.1] | 66 [44.8 to 70.3] | 46.5 [40.5 to 68]
Statistical Analysis 1: Comparison: Cont. Femoral Block - Low Dose Group vs Cont. Femoral Block - Higher Dose vs Continuous Adductor Canal; Test type: Superiority; p = 0.355, Kruskal-Wallis

2. Secondary Outcome: Average Length of Stay (to be Reported in Hours After Surgery)
Description: If pain is controlled and rehabilitation activity is optimal patient may be discharged at an earlier time
Time Frame: Participants will be followed for the duration of hospital stay; No patients will be discharged on the day of surgery; The earliest discharge would be at 24 hours. Those hospitalized beyond 96 hours will be excluded.
Measure: Median (Inter-Quartile Range); unit: Hours
Groups:
- Cont. Femoral Block - Low Dose Group: Arm is named by the intervention... Continuous Femoral Block - Low Dose. The Block/catheter is placed about 5cm below groin at ultrasonographic apex of femoral triangle. Rate of 2ml/hr of bupivacaine 0.0625% until morning of POD#2.
  Continuous Femoral Nerve Block: A 27g plastic catheter placed below the inguinal crease to perform a conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupi
- Cont. Femoral Block - Higher Dose: Place the CPNB in same manner as low-dose group, but rate will be 4ml/hr. Hypothesis is that this group may experience better pain control, but likely will have more motor blockade of thigh and less participation in physical therapy
  Continuous Femoral Nerve Block: A 27g plastic catheter placed below the inguinal crease to perform a conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupivacaine tho
Arm/Group | Cont. Femoral Block - Low Dose Group | Cont. Femoral Block - Higher Dose | Continuous Adductor Canal
Number analyzed (Participants) | 19 | 19 | 19
Hours | 75.5 [73 to 95.3] | 74.3 [70.3 to 80.8] | 72.5 [51.5 to 75.3]
Statistical Analysis 1: Comparison: Cont. Femoral Block - Low Dose Group vs Cont. Femoral Block - Higher Dose vs Continuous Adductor Canal; Test type: Superiority; p = 0.065, Kruskal-Wallis

3. Secondary Outcome: Postoperative Pain, Average Reported Score 11-point Scale
Description: The outcome is measured using a Numeric pain scale. The patient reports their average pain felt on postoperative day one, on a scale of 0 to 10 inclusive. Zero in this case indicates no pain at all and 10 indicates the worst pain they have ever felt.
Time Frame: postoperative day one
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Cont. Femoral Block - Low Dose Group | Cont. Femoral Block - Higher Dose | Continuous Adductor Canal
Number analyzed (Participants) | 19 | 19 | 19
units on scale | 3.961 (1.517) | 4.116 (1.638) | 4.282 (1.722)

4. Secondary Outcome: Sustained Straight Leg Raise
Description: Sustained Straight Leg Raise is the ability to elevate the heel and leg/knee off of bed for 5 seconds postoperatively after spinal anesthetic has resolved contralaterally.
Time Frame: Day of Surgery (DOS) - In Postoperative Recovery Unit, prior to any walking atempt
Measure: Count of Participants; unit: Participants
Arm/Group | Cont. Femoral Block - Low Dose Group | Cont. Femoral Block - Higher Dose | Continuous Adductor Canal
Number analyzed (Participants) | 19 | 19 | 19
Participants
  Yes | 19 | 14 | 16
  No | 0 | 1 | 0
  N/A | 0 | 4 | 3

ADVERSE EVENTS:
Time Frame: From enrollment on the day of surgery until discharge from the hospital, on average 3 days.
Groups:
- Cont. Femoral Block - Low Dose Group: Continuous Femoral Nerve Block (CFNB) -Low dose. The Block/catheter is placed about 5cm below groin usually corresponding with the ultrasonographic apex of femoral triangle. Rate of 2ml/hr of bupivacaine 0.0625% until morning of POD#2.
  CFNB: A 27g plastic catheter placed below the inguinal crease to perform a conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupivacaine is 0.0625%
- Cont. Femoral Block - Higher Dose: CFNB placed in same manner as low-dose group, but rate will be higher (4ml/hr). Hypothesis is this group may experience better pain control, but likely will have more motor blockade of thigh and less participation in physical therapy.
  CFNB: A 27g plastic catheter placed below the inguinal crease to perform a conduction blockade of the sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: The concentration of the continuous infusion of bupivacaine tho
- Continuous Adductor Canal: Placed at mid-thigh in proximal adductor canal near femoral artery with a bupivacaine infusion rate of 4ml/hr. Hypothesis is that this group may experience less motor blockade of thigh but may have more pain than the femoral nerve groups.
  Nerve Block, Continuous Adductor Canal: A 27g plastic catheter placed on the anterior-medial thigh midway between the Anterior Superior Iliac Spine (ASIS) and patella. Intent is to block sensory components of the femoral nerve in order to decrease pain in the knee after total knee arthroplasty.
  Continuous Sciatic Nerve Block: A transgluteal approach to the sciatic nerve is use to place a 27g catheter. It will only be dose postoperatively after verifying sciatic nerve function still intact. The infusion will be 0.003% bupivacaine at 2ml/hr. This is not the intervention of interest, but our institution's predominant practice is to include the sciatic nerve block as part of the analgesic regimen for total knee arthroplasty.
  Bupivacaine: T
Arm/Group | Cont. Femoral Block - Low Dose Group | Cont. Femoral Block - Higher Dose | Continuous Adductor Canal
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 1/21 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cont. Femoral Block - Low Dose Group (N=20) | Cont. Femoral Block - Higher Dose (N=21) | Continuous Adductor Canal (N=21)
Deep Vien Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes